CLINICAL TRIAL: NCT05795647
Title: The PENTO Protocol in Medication-related Osteonecrosis of the Jaw
Acronym: PENTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87RI21_0052 (PENTO)
Record Dates: First submitted 2022-12-14; First posted 2023-04-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Medication-related Osteonecrosis of the Jaw (MRONJ)
Keywords: MRONJ; pentoxifylline; tocophérol; bone exposure; renutrition
MeSH Terms: interventions — pentoxifylline-tocopherol-clodronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pentoxifylline (Experimental): Treatment will consist of pentoxifylline LP 400 mg morning and evening, combined with tocopherol 500 mg morning and evening
  Interventions: Drug: Pentoxifylline+Tocopherol

INTERVENTIONS:
Drug: Pentoxifylline+Tocopherol — Treatment will consist of pentoxifylline LP 400 mg morning and evening, combined with tocopherol 500 mg morning and evening

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) occurs after taking bisphosphonates or targeted therapies. It leads to a significant decrease in quality of life with pain, eating and chewing disorders, and malnutrition. Current treatments are only partially effective. PENTO (pentoxifylline and tocopherol) has been shown to be effective in maxillary osteoradionecrosis. The objective of this study is to evaluate the proportion of bone recovery in patients receiving PENTO in MRONJ at 12 months.

DETAILED DESCRIPTION:
MRONJ is defined as intraoral bone exposure persisting for more than 8 weeks after taking an anti-resorptive agent (per os or IV bisphosphonates, targeted therapies) and without history of maxilla radiotherapy or metastasis. It leads to a significant decrease in quality of life with significant pain at rest and during mastication, and compromised nutrition, sometimes resulting in severe undernutrition in patients already weakened by a history of cancer. Current treatments (prolonged antibiotic therapy, repeated bone curettage) have shown partial effectiveness. PENTO (combination of pentoxifylline, a vasodilator, and tocopherol, vitamin E) has been shown to significantly reduce intraoral exposed bone surface area and pain in maxilla osteoradionecrosis. All studies conducted so far on PENTO in MRONJ are retrospective or involve small samples. Therefore, our idea is to perform a well-conducted prospective phase IIa study to prove the efficacy of PENTO, with a larger sample size and identical follow-up periods. The investigators will study patients with AAOMS stage 2 MRONJ (exposed bone in symptomatic patients, without pathologic fracture).

Treatment will consist of pentoxifylline LP 400 mg morning and evening, combined with tocopherol 500 mg morning and evening. Antibiotic therapy with Augmentin (or clindamycin) will be added for the first month and then punctually if signs of local infection appear.

The primary and secondary endpoints will be assessed at inclusion and at 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Current or past treatment with bisphosphonates (oral or IV) and/or targeted therapies (denosumab, bevacizumab)
* Signs and symptoms for more than 8S with confirmation that the signs and symptoms are not of dental origin
* AAOMS Stage 2 MRONJ
* For patients of childbearing age, effective contraception is required

Exclusion Criteria:

* History of head or neck radiotherapy or maxilla metastases
* Patients who have received treatment in the past (PENTO or PENTOCLO protocol)
* Patients who have undergone surgery for their MRONJ within the last 3 months
* Pregnant or wishing to be pregnant, breastfeeding
* Patient under palliative care
* Patient with hypersensitivity to pentoxifylline or tocopherol or to an excipient
* History of hypersensitivity reaction to penicillins, cephalosporins, or other beta-lactams (and clindamycin or lincomycin if applicable) or excipient of amoxicillin-a. clavulanic or clindamycin
* History of jaundice/hepatic injury related to amoxicillin/clavulanic acid
* Patient taking oral anticoagulants, or with a history of major bleeding or bleeding disorders
* Patient taking platelet aggregation inhibitor, theophylline or aminophylline
* Patient taking methotrexate, probenecid, mycophenolate mofetil, myorelaxant drugs, macrolide or streptogramin antibiotics
* Patients with hepatic failure or renal failure (Cl < 30 mL/min),
* Patient with hypotension (SBP < 90 mmHg)
* Refusal to participate in the study
* Patient participating in other interventional research that may interfere with the conduct of this research
* Patient unable to understand the protocol
* Patient under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
Exposure bone area (EBA) | Month 12
  exposure bone area (EBA) less than 5 mm at 12 months. It will be expressed as the percentage of patients who achieved healing (EBA < 5 mm) at 12 months.

SECONDARY OUTCOMES:
SOMA score | Month 1, Month 3, Month 6, Month 12
  describe the evolution of the modified SOMA score (pain, chewing, bone exposure size, trismus, radiological appearance)
Nutritional parameters evolution (albuminemia) | Month 1, Month 3, Month 6, Month 12
  describe the nutritional parameters evolution albuminemia
Nutritional parameters evolution (pre-albuminemia) | Month 1, Month 3, Month 6, Month 12
  describe the nutritional parameters evolution pre-albuminemia
Nutritional parameters evolution (weight) | Month 1, Month 3, Month 6, Month 12
  describe the nutritional parameters evolution weight
Nutritional parameters evolution (BMI) | Month 1, Month 3, Month 6, Month 12
  describe the nutritional parameters evolution BMI
Exposure bone area (EBA) | Month 1, Month 3, Month 6, Month 12
  describe the evolution of the exposure bone area (EBA)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | Month 1, Month 3, Month 6, Month 12
  description of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Julie USSEGLIO, Dr, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges university hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No